CLINICAL TRIAL: NCT05797181
Title: The Effect of Medical Nutrition Therapy on Anthropometric Measurements and Blood Parameters in Sarcopenic Obesity Patients Receiving Peritoneal Dialysis Treatment
Brief Title: The Effect Of Medical Nutritional Therapy On Patients With Sarcopenic Obesity Receiving Peritoneal Dialysis Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Ayşe Betül Demirbaş, Principal Investigator, Atlas University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABDemirbasPD
Record Dates: First submitted 2023-02-24; First posted 2023-04-04 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Peritoneal Dialysis Complication; Sarcopenic Obesity
MeSH Terms: interventions — Nutrition Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary and Behavioral Change Group (Experimental): The experimental group will be required to adhere to a diet consisting of a 10-15% reduction in carbohydrate and a 1.2-1.4 g/kg body weight/day intake of protein.
  The participants will receive 4 times face-to-face meetings (on the first day and on week 1,5 and 9).
  Each face-to-face interview will last approximately 30 minutes. During the interview researcher will help the participants to determine their nutritional behaviors, plan and implement the diet.
  Interventions: Other: medical nutrition therapy in kidney diseases

INTERVENTIONS:
Other: medical nutrition therapy in kidney diseases — Planning and implementation of diets containing high protein, low potassium, low phosphorus, personalized adjusted carbohydrates

SUMMARY:
In this study, it was aimed to evaluate the effectiveness of medical nutrition therapy to be applied to patients with sarcopenic obesity receiving peritoneal dialysis treatment by measuring anthropometric measurements and blood parameters.

DETAILED DESCRIPTION:
Efficacy of medical nutrition therapy in patients with sarcopenic obesity receiving peritoneal dialysis treatment, general information form after patients filled in the voluntary consent form, SARC-F questionnaire as sarcopenia screening test, International Physical Activity Questionnaire (IPAQ), muscle mass, muscle strength, physical performance, BIA measurement, anthropometric measurements, laboratory findings and three-day food consumption records will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in research
* Be between the ages of 18-70
* To receive peritoneal dialysis treatment and to come to the hospital regularly once a month for treatment

Exclusion Criteria:

* Presence of any other disease that causes muscle wasting
* Patients using any supplement or enteral product in their diet

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Change in muscle strength | Baseline to 3 months after diet programme
  Handgrip strength (kg) will be measured by using the CAMRY EH101 dynamometer. Hand grip strength <16 kg for women and <27 kg for men indicates low muscle strength.
Change in the skeletal muscle mass | Baseline to 3 months after diet programme
  Skeletal muscle mass (kg) will be measured by using bioelectrical impedance analysis.
Change in the physical performance | Baseline to 3 months after diet programme
  4-meter walking speed test will be performed. A walking speed of ≤0.8 m/sec is considered as an indicator of severe sarcopenia.
Change of the fat mass | Baseline to 3 months after diet programme
  Fat mass (kg) will be measured by using bioelectrical impedance analysis.
Changes of percentage of body fat | Baseline to 3 months after diet programme
  Percentage of body fat will be measured by using bioelectrical impedance analysis.
Changes of body mass index | Baseline to 3 months after diet programme
  The weight and height will be combined to report BMI in kg/m2.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Betül Demirbaş, Principal Investigator — Atlas University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided